CLINICAL TRIAL: NCT00117546
Title: Cardiovascular Performance and Autonomic Reactivity in Formerly Preeclamptic Women With a Contracted Plasma Volume (CAPACITY Trial)
Brief Title: Cardiovascular and Autonomic Reactivity in Women With a History of Pre-eclampsia
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Radboud University Medical Center (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Diagnostic
Other Study IDs: 2004-155; P05.0007L
Record Dates: First submitted 2005-06-30; First posted 2005-07-07 (Estimated); Last update posted 2010-06-08 (Estimated); Status verified 2007-07

CONDITIONS: Preeclampsia
Keywords: CAPACITY trial; preeclampsia; plasma volume; sympathetic activity; hypertension; cardiovascular system
MeSH Terms: conditions — Pre-Eclampsia; Hypertension | interventions — Methyldopa

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: alpha methyldopa — 500 mg twice a day
  Other Names: Aldomet

SUMMARY:
A history of preeclampsia is associated with a low plasma volume and higher sympathetic activity. Methyldopa will suppress sympathetic activity to normal values. In this study, the researchers will test that effect on the total cardiovascular balance.

DETAILED DESCRIPTION:
This is a randomized double-blind placebo controlled cross-over study in formerly preeclamptic women with a contracted plasma volume. The researchers will test the effect of methyldopa on the cardiovascular balance and orthostatic tolerance in women with a history of preeclampsia and healthy controls.

ELIGIBILITY:
Inclusion Criteria:

* Primiparous
* History of preeclampsia
* Low plasma volume

Exclusion Criteria:

* Thrombophilia
* Hypertension
* Auto-immune disorder
* Insulin dependent diabetes mellitus

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2005-09; Study Completion 2008-12 (Estimated)

PRIMARY OUTCOMES:
normalized plasma volume | 1 month

SECONDARY OUTCOMES:
increased orthostatic tolerance | 1 month
normalized cardiovascular balance | 1 month
venous capacitance | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Ineke Krabbendam, MD, Principal Investigator — Department of Obstetrics and Gynaecology, Radboud University Nijmegen Medical Centre
Locations (1):
- Radboud University Nijmegen Medical Center, Nijmegen, Netherlands